CLINICAL TRIAL: NCT03797118
Title: The First Experience With Using a One-dimensional Mathematical Model With Fully Automated Algorithm of Extraction of Patient-specific Geometry From CT Images for a Noninvasive Assessment of Fractional Flow Reserve.
Brief Title: One-Dimensional Mathematical Model-Based Automated Assessment of Fractional Flow Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Daria Gognieva, Principal Investigator, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-51-53160
Record Dates: First submitted 2018-12-22; First posted 2019-01-08 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease
Keywords: noninvasive assessment of the fractional flow reserve; coronary computed tomography angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FFRct (Experimental): Patients will receive cCTA, ICA, FFRct, and FFRinv per protocol.
  Interventions: Device: FFR

INTERVENTIONS:
Device: FFR — Fractional flow reserve measured during cardiac catheterization

SUMMARY:
This study evaluates the diagnostic efficiency of an automated method of noninvasive assessment of the fractional reserve of coronary blood flow.

Fractional flow reserve is estimated with a one-dimensional mathematical model constructed by means of an automated algorithm. Noninvasive method values are thereafter compared with invasive method values.

DETAILED DESCRIPTION:
Noninvasive assessment of Fractional Flow Reserve is almost never applied in the Russian Federation due to the relative novelty and study insufficiency, lack of the appropriate resource base, specific necessary software and trained qualified personnel.

In 2015, scientists from the Institute of Numerical Mathematics RAS in collaboration with specialists of the I.M. Sechenov First Moscow State Medical University developed a noninvasive method of fractional flow reserve assessment based on a one-dimensional mathematical model. A model is constructed based on images derived from the coronary computed tomography angiography performed by standard protocol; the method is fully automated.

The aim of our study is to evaluate the diagnostic efficiency of this technique in clinical practice.

This is a pilot study; we are planning to enroll 30 patients: 13 of them underwent 64-slice computed tomography and are included retrospectively; 17 will be included prospectively, with a 640-slice CT scan. Specialists from the Laboratory of Mathematical Modeling will process CT images and evaluate noninvasive FFR. Ischemia is confirmed if FFR < 0.80 and disproved if FFR ≥ 0.80. After that, the prospective group of patients will be hospitalized for invasive FFR assessment as a reference standard; if ischemia is proved, patients will undergo stent implantation. In the retrospective group, patients already have invasive FFR values estimated.

Statistical analysis will be performed using R programming language packages (cran-r.project.com). Continuous variables will be presented as mean values ± standard deviations, order variables will be presented as medians with interquartile ranges in parentheses. We are going to use the D'Agostino-Pearson omnibus test for the assessment of normality of distribution and construct a Q-Q Plot. We will compare these two methods with the Bland-Altman analysis and ROC-analysis and will assess the degree of correlation with the Pearson's chi-squared.

The study should result in determining the sensitivity, specificity, positive and negative predictive values of the method.

After the active phase of the research is done, we are planning to proceed observation on the prospective group of patients to verify the endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients providing written informed consent
2. Scheduled to undergo clinically-indicated non-emergent invasive coronary angiography (ICA)
3. Has undergone >640 multidetector CCTA within 60 days prior to ICA
4. No cardiac interventional therapy between the CCTA and ICA

Exclusion Criteria:

1. Prior coronary artery bypass graft (CABG) surgery
2. Prior percutaneous coronary intervention (PCI) for which suspected coronary artery lesion(s) are within a stented coronary vessel
3. Contraindication to adenosine, including 2nd or 3rd-degree heart block; sick sinus syndrome; long QT syndrome; severe hypotension, severe asthma, severe COPD or bronchodilator-dependent COPD
4. Suspicion of acute coronary syndrome (acute myocardial infarction and unstable angina)
5. Recent prior myocardial infarction within 40 days of ICA
6. Known complex congenital heart disease
7. Prior pacemaker or internal defibrillator lead implantation
8. Prosthetic heart valve
9. Significant arrhythmia or tachycardia
10. Impaired chronic renal function (serum creatinine >1.5 mg/dl
11. Patients with known anaphylactic allergy to iodinated contrast
12. Pregnancy or unknown pregnancy status
13. Body mass index >35
14. Patient requires an emergent procedure
15. Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema
16. Any active, serious, life-threatening disease with a life expectancy of less than 2 months
17. Inability to comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of FFRct | through study completion, an average of 8 months
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of FFRct at the vessel level using binary outcomes whith compared to FFR as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Daria Gognieva, MD, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University); Philipp Kopylov, Professor, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Daria Gognieva, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Data disclosure is not permitted by the local ethics committee. For more information about the study, you need to contact the principal investigator.

REFERENCES:
- [Background] Gognieva D, Gamilov T, Pryamonosov R, Betelin V, Ternovoy SK, Serova NS, Abugov S, Shchekochikhin D, Mitina Y, El-Manaa H, Kopylov P. One-Dimensional Mathematical Model-Based Automated Assessment of Fractional Flow Reserve in a Patient with Silent Myocardial Ischemia. Am J Case Rep. 2018 Jun 20;19:724-728. doi: 10.12659/AJCR.908449. PMID 29921835
- See also: Am J Case Rep. 2018 Jun 20;19:724-728. doi: 10.12659/AJCR.908449. — https://www.ncbi.nlm.nih.gov/pubmed?term=Am+J+Case+Rep+%5BJour%5D+AND+One-Dimensional+Mathematical+Model-Based+Automated+Assessment+of+Fractional+Flow+Reserve+in+a+Patient+with+Silent+Myocardial+Ischemia&TransSchema=title&cmd=detailssearch